CLINICAL TRIAL: NCT00285246
Title: Prospective Study of Functional Status in Veterans at Risk for Unexplained Illnesses
Brief Title: Prospective Study of Veteran Health in Previously Deployed Soldiers
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 02-296
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Combat Disorders
Keywords: combat disorders; stress, psychological; somatoform disorders; life change events; utilization
MeSH Terms: conditions — Combat Disorders; Stress, Psychological; Somatoform Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Army Reserve and National Guard soldiers deploying to a hazardous deployment from Fort Dix, NJ and Camp Shelby, MS

SUMMARY:
Background: Previous deployments like that to the Persian Gulf in 1991 produced veterans with post-deployment symptom-based health problems with no medical explanation. This was termed Gulf War illness or medically unexplained illness (MUI). If previous wars are any indication, some soldiers currently deployed to hostile areas also will return home with unexplained symptom-based illnesses. However, when this study began there was virtually no pre-war, prospective data on risk and resilience factors associated with MUI. This study is attempting to fill that gap.

Objectives: Our goals are to: (a) determine pre- and immediate post-deployment factors predicting later MUI and poor functional status, (b) improve previous methodological problems (e.g., selection bias, recall bias and lack of baseline controls) in studies of MUI, and (c) relate pre-deployment risk factors (e.g., personality, stressor reactivity) and resilience factors (e.g., coping style, social support) to post-deployment functional status.

DETAILED DESCRIPTION:
Background: Previous deployments like that to the Persian Gulf in 1991 produced veterans with post-deployment symptom-based health problems with no medical explanation. This was termed Gulf War illness or medically unexplained illness (MUI). If previous wars are any indication, some soldiers currently deployed to hostile areas also will return home with unexplained symptom-based illnesses. However, was virtually no pre-war, prospective data on risk and resilience factors associated with MUI before 2001. This study will attempt to fill that gap. Objectives: Our goals are to: (a) determine pre- and immediate post-deployment factors predicting later MUI and poor functional status, (b) improve previous methodological problems (e.g., selection bias, recall bias and lack of baseline controls) in studies of MUI, and (c) relate pre-deployment risk factors (e.g., personality, stressor reactivity) and resilience factors (e.g., coping style, social support) to post-deployment functional status. Methods: This study uses a prospective, longitudinal observational design to assess risk and resilience factors for post-war MUI in Reserve and National Guard enlisted personnel. A stratified random sample of more than 700 subjects will be drawn from those undergoing pre- and post-mobilization readiness processing at Fort Dix, NJ and Camp Shelby, MS. Personnel will be tested pre-mobilization (Phase 1), immediately after mobilization (Phase 2) and at 3 months and 1 year post-deployment (Phases 3 & 4). Predictor variables include personality, social support, coping style, non-specific symptoms, sympathetic cardiac stress reactivity, and cortisol stress reactivity. Control variables include prior traumatic events, current distress, PTSD symptoms, socially desirable responding, body mass index, deployment experiences, environmental exposures and demographics (e.g., age, gender). Outcome variables include functional status, healthcare utilization, and MUI status (using CDC criteria for chronic multisymptom illness developed after the first Gulf War). Status: Publications and presentations are being prepared. Impact: The larger, prospective study with soldiers will help us to identify pre- and early post-deployment risk and resilience factors important in MUI, functional status, and healthcare utilization. There is an urgent need for both pre- and post-deployment predictors of later MUI uncontaminated by recall bias, and the selection bias of studying only treatment-seekers. If we are to understand how to best treat veterans presenting with unexplained symptoms, then we need to know which pre-war factors are most useful in predicting who is most likely to be resilient and who is most likely to be at risk for later unexplained illness.

ELIGIBILITY:
Inclusion Criteria:

* Army Reserve and National Guard soldiers deploying to a hazardous deployment from Fort Dix, New Jersey (NJ) and Camp Shelby, Mississippi (MS)

Exclusion Criteria:

* There are some drug exclusions for anything that substantially affects cardiovascular function.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Army National Guard & Reserves Soldiers deploying to either Iraq or Afghanistan. Outcome measures assessed at all 4 time points (pre-deployment, immediately post-deployment, 3 months post-return, 1 year post-return)
Sampling Method: Non-Probability Sample
Enrollment: 838 (Actual)
Dates: Start 2005-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen S. Quigley, PhD, Principal Investigator — East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ
Locations (2):
- United States (2):
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey

REFERENCES:
- [Result] McAndrew LM, D'Andrea E, Lu SE, Abbi B, Yan GW, Engel C, Quigley KS. What pre-deployment and early post-deployment factors predict health function after combat deployment?: a prospective longitudinal study of Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) soldiers. Health Qual Life Outcomes. 2013 Apr 30;11:73. doi: 10.1186/1477-7525-11-73. PMID 23631419
- [Result] Yan GW, McAndrew L, D'Andrea EA, Lange G, Santos SL, Engel CC, Quigley KS. Self-reported stressors of National Guard women veterans before and after deployment: the relevance of interpersonal relationships. J Gen Intern Med. 2013 Jul;28 Suppl 2(Suppl 2):S549-55. doi: 10.1007/s11606-012-2247-6. PMID 23807064
- [Result] Falvo MJ, Serrador JM, McAndrew LM, Chandler HK, Lu SE, Quigley KS. A retrospective cohort study of U.S. service members returning from Afghanistan and Iraq: is physical health worsening over time? BMC Public Health. 2012 Dec 28;12:1124. doi: 10.1186/1471-2458-12-1124. PMID 23272950
- [Result] Quigley KS, McAndrew LM, Almeida L, D'Andrea EA, Engel CC, Hamtil H, Ackerman AJ. Prevalence of environmental and other military exposure concerns in Operation Enduring Freedom and Operation Iraqi Freedom veterans. J Occup Environ Med. 2012 Jun;54(6):659-64. doi: 10.1097/JOM.0b013e3182570506. PMID 22588478

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Army Reserve and National Guard soldiers deploying to a hazardous deployment from Fort Dix, NJ and Camp Shelby, MS
Period: Overall Study
Arm/Group | All Participants
Started | 838
Completed | 790 (Number of participants who were eligible and completed at least one phase of data collection)
Not Completed | 48

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | All Participants
Number analyzed (Participants) | 838
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 742
Race/Ethnicity, Customized [Number; unit: participants]
  White/Causasian | 564
  Hispanic/Latino | 33
  Black/African American/Non-Hispanic | 72
  Black/African American/Hispanic | 1
  Asian | 12
  Native Hawaiian or other Pacific Islander | 10
  American Indian or Alaskan Native | 46
  Unknown/Not Provided | 100
Region of Enrollment [Number; unit: participants]
  United States | 838

OUTCOME MEASURES:

1. Primary Outcome: Non-Specific Physical Symptoms
Description: Severity of non-specific physical symptoms from the 15 item Patient Health Questionnaire-15 (Kroenke, Spitzer & Williams, 2002). Scale score range is 0-30. Higher scores indicate greater non-specific physical symptom severity. This scale does not contain subscales.
Time Frame: pre-deployment (Phase 1), immediately post-deployment (Phase 2), 3 months post-return from deployment (Phase 3), 1 year post-return from deployment (Phase 4)
Population: Not all of the 790 completers has complete data on the non-specific physical symptoms measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 767
units on a scale
  Phase 1 | 5.2 (3.9)
  Phase 2 | 7.9 (4.9)
  Phase 3 | 7.7 (5.1)
  Phase 4 | 7.7 (5.4)

2. Primary Outcome: Physical Functional Status
Description: Physical Component Summary Score (PCS) from the Veterans RAND (VR) 36 measure (Kazis, 2000). Composite scores are normed to a mean of 50 and a SD of 10. Scores can range from 0-100. Higher scores indicate better physical function.
Time Frame: pre-deployment (Phase 1), immediate post-deployment (Phase 2), 3 months post-return (Phase 3), 1 year post-return (Phase 4)
Population: Not all of the 790 completers has complete data on this physical functional status measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 762
Units on a scale
  Phase 1 | 55.5 (5.2)
  Phase 2 | 53.7 (6.9)
  Phase 3 | 52.8 (7.6)
  Phase 4 | 51.5 (8.8)

3. Primary Outcome: Mental Functional Status
Description: Mental Component Summary Score (MCS) from the Veterans-RAND (VR) 36 (Kazis, 2000). MCS is a composite score with a mean of 50 and a standard deviation of 10. Scale scores range from 0-100 with higher scores reflecting better mental function.
Time Frame: pre-deployment, immediate post-deployment, 3 months post-return, 1 year post-return
Population: Not all of the 790 completers has complete data on the mental functional status measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 762
units on a scale
  Phase 1 | 48.0 (9.1)
  Phase 2 | 45.7 (10.7)
  Phase 3 | 45.0 (11.5)
  Phase 4 | 44.9 (12.4)

4. Primary Outcome: Health Care Utilization
Description: This variable is a sum score of the self-reported number of healthcare provider visits and emergency room visits in the prior 12 months.
Time Frame: as for outcome 2
Population: Not all of the 790 completers has complete data on the healthcare utilization measure.
Measure: Mean (Standard Deviation); unit: number of visits in prior 12 months
Arm/Group | All Participants
Number analyzed (Participants) | 752
number of visits in prior 12 months
  Phase 1 | 0.78 (0.87)
  Phase 2 | 0.68 (0.81)
  Phase 3 | 0.69 (0.74)
  Phase 4 | 1.11 (0.97)

ADVERSE EVENTS:
Time Frame: Data were collected at all 4 time points (pre-deployment=Phase 1, immediate post-deployment=Phase 2, 3 months post-deployment=Phase 3, one year post-deployment=Phase 4). The entire duration was about 2 years given an average deployment of about one year.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/838
Other Adverse Events (participants affected / at risk) | 0/838

LIMITATIONS AND CAVEATS:
The sample was comprised of only Army National Guard and Reserve military personnel, and therefore results may not generalize to the broader population of military personnel from other Service branches or components.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes